CLINICAL TRIAL: NCT02387450
Title: Reduction de la Morbi-mortalité Cardiovasculaire Chez l'artériopathe Claudicant Par le Sildenafil
Brief Title: Reduced Cardiovascular Morbi-mortality by Sildenafil in Patients With Arterial Claudication
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ongoing recording
Record Dates: First submitted 2015-03-02; First posted 2015-03-13 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Peripheral Arterial Disease
Keywords: Claudication; Maximal walking distance; Morbi-mortality
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treated group (Active Comparator): Sildenafil, oral, 100mg per day
  Interventions: Drug: Sildenafil
- Control group (Placebo Comparator): placebo oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — 100 mg per day
  Other Names: Viagra or revatio
  Arms: Treated group
Drug: Placebo — Placebo with same presentation as the active drug
  Arms: Control group

SUMMARY:
Sildenafil has shown potential effects both on vasodilator mechanisms and as an inhibitor of the NO/GMPc Pain activation. The investigators aim at estimating the benefit of sildenafil in term of morbi-mortality in patients with arterial claudication on a multicenter prospective double blind study.

DETAILED DESCRIPTION:
Eligible patients will ask to participate after oral and written information. Evaluation of walking capacity (self reported and treadmill measured), co-morbid condition and quality of life (WELCH, SF-36, Edinburg) will be performed at inclusion, after the first dose and at 3 months of oral treatment through sildenafil 100mg/day or placebo from inclusion to 3 months.

Indication for revascularisation will be evaluated at 3 months according to symptoms and walking capacity according to the Rutherford classification.

Primary endpoint is the proportion of patients showing either a fatal events (cardio-vascular or noncardiovascular) or hospitalisation for non fatal cardiovascular events at 6 and 9 months follow up from inclusion.

ELIGIBILITY:
Inclusion Criteria:

* ABI<0.90
* Vascular type claudication
* stable walking impairment for at least 3 months
* Optimal cardiovasc treatment (Anti-platelet, HMGCoA-Inh, ACE-Inh or AT2 inh)
* Age > 30 years

Exclusion Criteria:

* Refuse to participate
* Administrative protection
* Severe renal (clearance < 30 ml/min) or hepatic (Child-Pugh C) failure

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Morbi-mortality : combined criterion (Cardiovascular fatal and non fatal event Improvement of 1 stage) | 6 months

SECONDARY OUTCOMES:
Quality of life Questionnaire | 3, 6 and 9 months
Safety and secondary effects (Headache, Hypotension) (Proportion of Participants with Adverse Event) | 3, 6 and 9 months
  Proportion of Participants with Adverse Events (sildenafil vs. placebo)
Walking capacity (treadmill test) | 3, 6 and 9 months
  treadmill test
Proportion of revascularized patients | 6 and 9 months
  Revascularisation

CONTACTS AND LOCATIONS:
Overall Officials: pierre Abraham, MD, PhD, Principal Investigator — University Hospital in Angers
Locations (1):
- Centre hospitalier universitaire, Angers, France